CLINICAL TRIAL: NCT01606566
Title: Open-label, Single Arm, Multi-centre, Phase II Study to Evaluate the Safety and Efficacy of Amphinex Induced PCI of Bleomycin With Superficial and Interstitial Laser Light Application in Patients With Recurrent Head and Neck Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Amphinex Induced PCI of Bleomycin for Recurrent Head and Neck Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: PCI Biotech AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCIA202/10; 2011-003751-19 (EudraCT Number)
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Head and Neck Cancer; Carcinoma, Squamous Cell of Head and Neck
Keywords: Recurrent; Head and Neck; Neoplasms; Squamous Cell Carcinoma; Amphinex; Cancer; Photodynamic therapy; Chemotherapy; Bleomycin
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasms; Carcinoma, Squamous Cell | interventions — Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amphinex induced PCI of bleomycin (Experimental): Drug: Amphinex induced PCI of bleomycin
  Intervention:Intravenous administration of Amphinex (day 0) followed by intravenous administration of bleomycin and laser light application (day 4). Laser light application could be both interstitial and/or superficial depending on the tumour location.
  Interventions: Drug: Amphinex induced PCI of bleomycin

INTERVENTIONS:
Drug: Amphinex induced PCI of bleomycin — Intravenous administration of 0.25 mg/kg Amphinex (day 0) followed by intravenous administration of bleomycin (15000 IU/m2, day 4) and laser light application (3 hours (+/- 1 hour) after bleomycin administration).
  Other Names: Blenoxane

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Amphinex induced PCI of bleomycin ('PC-A11') with superficial and/or interstitial laser light application in patients with recurrent SCCHN.

DETAILED DESCRIPTION:
Approximately 650 000 new cases of head and neck cancer are diagnosed worldwide each year (2). Europe alone, it is estimated that there are approximately 143 000 new cases and more than 68 000 deaths each year (3). The vast majority (>90%) of head and neck malignancies are squamous cell carcinomas. Most (60-70%) patients with squamous cell carcinoma of the head and neck (SCCHN) present with loco regionally advanced disease.

Standard treatment options for SCCHN include surgery, radiotherapy and chemotherapy. Single-modality treatment with surgery or radiotherapy is generally recommended for the 40% of patients who present stage I or II disease. Each of the two modalities results in similar survival with cure rates ranging between 60% and 90%.

For the 60% of the patients who present with locally advanced disease at diagnosis, combined modality therapy is generally recommended. For patients with unresectable disease the current standard treatment is concurrent cisplatin-based chemoradiation. This is also the standard for patients with resectable disease when organ preservation is desired and, as adjuvant treatment, for patients with high-risk pathological findings at surgical resection.

Despite such an approach, a substantial percentage of patients (20-30%) develop local and/or regional recurrences and distant metastases. Recurrent disease is often not resectable, and even in resectable cases, some patients decline the surgical procedure due to quality of life considerations. Additionally, in recurrent disease the radiation tolerance of the normal tissues makes re-irradiation technically challenging and frequently more toxic than the initial course. The prognosis of patients with recurrent or metastatic SCCHN is generally poor, with a median survival of 6-9 months.

The therapeutic ratio in recurrent SCCHN is narrow. Therefore, there is a large unmet medical need for novel treatments in this patient group, both to lengthen overall survival, and to improve the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Study eligibility reviewed and approved by interdisciplinary hospital team.
2. Age minimum 18 years.
3. Histologically or cytological confirmed diagnosis of recurrent or metastatic SCCHN considered unsuitable for surgery and radiotherapy (patients with distant or regional metastatic disease may be eligible if local palliation is needed)
4. Performance status (WHO scale/ECOG) ≤ 1.
5. At least one measurable target lesion at baseline.
6. Local disease including margin (0.5 cm) treatable with superficial and/or interstitial laser light application (for superficial lesions: entire tumour assessable for laser light application/interstitial treatment: insertion of implants feasible)
7. Estimated life expectancy of at least 12 weeks.
8. Written informed consent.

Exclusion criteria:

Prior Treatment:

1. Local treatment of their SCCHN by surgery within the previous 4 weeks or by radiation within the previous 3 months.
2. Previous treatment with systemic chemotherapy for their SCCHN within the last 4 weeks
3. Previous treatment with Photodynamic Therapy within the last 6 months.
4. Prior treatment with bleomycin.
5. Prior treatment with PC-A11.
6. Toxicities incurred as a result of previous anticancer therapy (radiation therapy, chemotherapy, or surgery) which did not resolve to ≤ grade 2.

   Current Treatment:
7. Current or recent (within 30 days of first study treatment) treatment with another investigational drug or participation in another investigational study.
8. Other concurrent anticancer therapies.
9. Treatment with a medicinal product with known or potential drug-drug interaction with bleomycin or Amphinex.

   Haematology, coagulation and biochemistry:
10. Inadequate bone marrow function:

    Absolute Neutrophil Count (ANC): < 1.5 x 109/L, or platelet count <100 x 109/L or haemoglobin < 6 mmol/L.
11. Inadequate liver function, defined as:

    Serum (total) bilirubin > 2 x the Upper Limit of Normal (ULN) for the institution.

    Aspartate Amino Transferase (ASAT) or Alanine Amino Transferase (ALAT) > 2.5 x ULN.

    Alkaline phosphatase levels > 2.5 x ULN.
12. Glomerular filtration rate (GFR) < 30ml/min.
13. Clinical significant electrolyte abnormalities (Potassium, Magnesium, Phosphate that is greater than CTCAE grade 3 for both low and high values)

    Other:
14. Tumours known or suspected to be eroding into a major blood vessel, e.g. carotid artery (interna and /or communis) in or adjacent to the illumination site (minimum distance between tumour tissue and critical structure should be 0.5 cm).
15. Nasopharyngeal carcinoma.
16. Conditions contraindicated for bleomycin treatment (current lung infection, severely impaired pulmonary function) excluded by lung function test (either formal lung function test for patients able to undertake such assessment, or a suitable opinion by an appropriately trained Respiratory / Anaesthetic Clinical Specialist).
17. Conditions that worsen when exposed to light (including porphyria).
18. Inability to undergo CT or MRI.
19. Pregnancy or lactation (female patients with childbearing potential). Serum pregnancy test to be performed within 7 days prior to study PC-A11 treatment start, or within 14 days followed by a confirmatory urine pregnancy test within 7 days prior to study treatment start.
20. For female patients of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male patients who are not surgically sterile or with female partners of childbearing potential: absence of highly effective method of contraception resulting in a low failure rate (i.e. less than 1% per year). These methods of contraception according to the note for guidance on non-clinical safety studies for the conduct of human trials for pharmaceuticals (CPMP/ICH/286/95, modification) include consistent and correct use of hormone containing implants and injectables, combined oral contraceptives, hormone containing intrauterine devices, surgical sterilization, sexual abstinence and vasectomy. Note: Abstinence is only acceptable as true abstinence: when this is in line with the preferred and usual lifestyle of the subject, periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
21. Planned surgery, endoscopic examination or dental treatment in first 30 days after PC-A11 treatment.
22. Co-existing ophthalmic disease likely to require slit-lamp examination within the first 90 days after PC-A11 treatment.
23. Congestive heart failure New York Heart Association (NYHA) Class III and IV. Cardiac arrhythmias (except for atrioventricular block type I, Mobitz type II, and Wenckebach type) signs and symptoms of relevant cardiovascular disease.
24. Known allergy or sensitivity to photosensitisers.
25. Ataxia telangiectasia
26. Concomitant malignant disease, with exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix.
27. Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, physical examination or laboratory findings) that may interfere with the planned PC-A11 treatment, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-04; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | 3 months
  The 'run-in part' primary endpoint
The proportion of patients with non-progressive local disease at 6 months | 6 months
  The expansion part primary endpoint

SECONDARY OUTCOMES:
Pharmacokinetics of 'PC-A11' in plasma | 3 months
  The run-in part and expansion part secondary endpoint
The proportion of patients with non-progressive local disease at 3 months | 12 months
  The run-in part and expansion part secondary endpoint
Proportion of patients with adverse events | 12 months
  The run-in part and expansion part safety endpoint
Progression free survival | 12 months
  The run-in part and expansion part secondary outcome measure
QoL using EORTC Quality of Life Questionnaire (QLQ)-C30 version 3.0 and QLQ-H&N35 | 12 months
  The run-in part and expansion part secondary outcome measures

OTHER OUTCOMES:
Evaluation of biomarkers obtained from tumour tissue and blood samples | 12 months
  The run-in part and expansion part secondary outcome measure
Evaluation of skin photosensitivity | 3 months
  The run-in part and expansion part secondary outcome measure
Evaluation of local tumour responses by volumetric measurements. | 12 months
  The run-in part and expansion part secondary outcome measure
Evaluation of fluorescence of tumour tissue | Day 4
  The run-in part and expansion part secondary outcome measure
Evaluation of pain | 12 months
  Scored by a visual analogue score (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Baris Karakullukcu, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (10):
- France (2):
  - CHU de Nantes Hôtel Dieu, Nantes, Nantes Cedex 1
  - Centre Alexis Vautrin (CAV)-Nancy Université, Nancy
- Germany (4):
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Charité Comprehensive Cancer Center, Berlin
  - Universitätsklinikum Essen, Essen
  - Ludwig Maximilian University Munich, München
- Institute of Oncology, Vilnius University, Vilnius, Lithuania
- The Netherlands Cancer Institute, Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands
- Szpital Specjalistyczny w Brzozowie, Brzozów, Poland
- University College London Hospital, London, United Kingdom

REFERENCES:
- See also: Click here to for more information about the Sponsor of the study — http://www.pcibiotech.no